CLINICAL TRIAL: NCT00925795
Title: Effect of Extra Virgin Olive Oil on Atherosclerosis Biomarkers in Patients Treated With Combination Antiretroviral Therapy: a Randomized, Crossover Trial
Brief Title: Effect of Extra Virgin Olive Oil on Atherosclerosis Biomarkers in HIV-infected Patients
Acronym: EVOO_HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Josip Begovac, MD, PhD, professor in infectious diseases, University Hospital for Infectious Diseases "Dr Fran Mihaljevic"
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UHID-01
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: HIV; Atherosclerosis; HIV Infections
Keywords: HIV; atherosclerosis; extra virgin olive oil; Alternative therapies; Treatment experienced+
MeSH Terms: conditions — Atherosclerosis; HIV Infections | interventions — Economics; Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (1. EVOO; 2. ROO) (Active Comparator)
  Interventions: Other: consumption 1. EVOO; 2. ROO
- Group B (1. ROO; 2. EVOO) (Active Comparator)
  Interventions: Other: consumption 1. ROO; 2. EVOO

INTERVENTIONS:
Other: consumption 1. EVOO; 2. ROO — EVOO in doses of 50 mL/daily for 20 days; 14 days of wash-out period without olives and olive oil; followed by ROO in doses of 50 mL/daily for 20 days
  Other Names: olive oil
  Arms: Group A (1. EVOO; 2. ROO)
Other: consumption 1. ROO; 2. EVOO — ROO in doses of 50 mL/daily for 20 days; 14 days of wash-out period without olives and olive oil; followed by EVOO in doses of 50 mL/daily for 20 days
  Other Names: olive oil
  Arms: Group B (1. ROO; 2. EVOO)

SUMMARY:
HIV infection is associated with systemic inflammation that is involved in pathogenesis of atherosclerosis. Treatment of HIV infection may cause lipid profile disturbance and consequently, atherosclerosis progression. In general, extra virgin olive oil (EVOO) has beneficial effect on atherosclerosis markers. Our goals are to examine the effect of EVOO on atherosclerosis markers in HIV-treated patients. A controlled randomized cross-over study will be performed on 40 participants. They will consume EVOO and ROO (refined olive oil) during two 20 days intervention periods, interrupted with 14 days wash-out period. Before the trial and after both intervention periods we will analyze participants' blood for: ESR, white blood cell count, hsCRP, interleukin-6, oxidized LDL, glutathione peroxidase, superoxide dismutase, malondialdehyde, triglycerides, total cholesterol, HDL and LDL cholesterol, fibrinogen, factor VII and von Willebrand factor. We expect an improvement of these parameters after three weeks of EVOO consumption.

DETAILED DESCRIPTION:
There are many studies about beneficial effect of extra virgin olive oil on atherosclerosis biomarkers. Our study investigates the same, but in population of HIV-infected patients receiving antiretroviral treatment. The main health benefit of EVOO can be attributed to high content of phenolic compounds, that have a favorable effect on blood pressure, LDL oxidation, platelet aggregation, endothelial function, oxidative stress. We analyzed the total phenolic compounds (PC) in different types of olive oils and decided to use EVOO with four times higher levels of PC than refined olive oil (ROO) which we would use as placebo.

A randomized crossover controlled trial will be performed on 40 participants with signed informed consent. They will be randomly divided in two groups. Each group will consume two types of olive oils (EVOO and ROO) in two intervention periods, but in different order. That means that group "A" will consume EVOO in the first and ROO in the second intervention period. Group "B" has inversed order of olive oil administration. Two intervention periods of 20 days will be interrupted with wash-out period of 14 days. During intervention periods participants will consume daily doses of 50 mL of particular olive oil. During wash-out periods participants should avoid olives and olive oil consumption. Before the first and after each of the two intervention periods, blood will be taken. Some of the tests will be done immediately after blood sample collection (glucose, hsCRP, triglycerides, total cholesterol, HDL and LDL cholesterol, CBC, ESR). For some of the tests (IL-6, von Willebrand factor, factor VII, oxidated LDL, glutathione peroxidase, superoxide dismutase) the specimens will be collected and stored at -80°C until the analysis.

As many studies showed improvement of these parameters in population affected with atherosclerosis, we could also expect the similar effect in HIV-infected patients who are more likely to develop atherosclerosis, partly because of HIV-infection itself and partly because of side effects of antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive patients receiving antiretroviral drugs
* undetectable HIV viral load in plasma for at least 6 months (by high sensitive Amplicor HIV-1 Monitor, version 1.5)
* glucose level within reference range

Exclusion Criteria:

* pregnant HIV-positive women
* HIV-patients with underlying acute/chronic diseases (except cardiovascular)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To assess whether consumption of extra virgin olive oil (EVOO) leads to improvement of atherosclerosis biomarkers in persons receiving antiretroviral drugs. | biomarker measurement before and after both intervention periods (20 days each)

SECONDARY OUTCOMES:
To assess which atherosclerosis biomarkers are the most affected (inflammation, hypercoagulability, dislipidemia, endothelial dysfunction or oxidative stress) by EVOO consumption | biomarker measurement before and after both intervention periods (20 days each)

CONTACTS AND LOCATIONS:
Overall Officials: Josip Begovac, MD, PhD, Principal Investigator — University Hospital for Infectious Diseases "Dr Fran Mihaljevic" Zagreb, Croatia
Locations (1):
- University Hospital for Infectious Diseases "Dr Fran Mihaljevic", Zagreb, Croatia

REFERENCES:
- [Background] Covas MI. Olive oil and the cardiovascular system. Pharmacol Res. 2007 Mar;55(3):175-86. doi: 10.1016/j.phrs.2007.01.010. Epub 2007 Jan 30. PMID 17321749
- [Background] Perona JS, Cabello-Moruno R, Ruiz-Gutierrez V. The role of virgin olive oil components in the modulation of endothelial function. J Nutr Biochem. 2006 Jul;17(7):429-45. doi: 10.1016/j.jnutbio.2005.11.007. Epub 2005 Dec 12. PMID 16481154
- [Background] Covas MI, Nyyssonen K, Poulsen HE, Kaikkonen J, Zunft HJ, Kiesewetter H, Gaddi A, de la Torre R, Mursu J, Baumler H, Nascetti S, Salonen JT, Fito M, Virtanen J, Marrugat J; EUROLIVE Study Group. The effect of polyphenols in olive oil on heart disease risk factors: a randomized trial. Ann Intern Med. 2006 Sep 5;145(5):333-41. doi: 10.7326/0003-4819-145-5-200609050-00006. PMID 16954359
- [Background] Mehta N, Reilly M. Atherosclerotic cardiovascular disease risk in the HAART-treated HIV-1 population. HIV Clin Trials. 2005 Jan-Feb;6(1):5-24. doi: 10.1310/HT0W-NX2N-U2BM-7LUU. PMID 15765307
- [Background] Francisci D, Giannini S, Baldelli F, Leone M, Belfiori B, Guglielmini G, Malincarne L, Gresele P. HIV type 1 infection, and not short-term HAART, induces endothelial dysfunction. AIDS. 2009 Mar 13;23(5):589-96. doi: 10.1097/QAD.0b013e328325a87c. PMID 19177019
- [Derived] Kozic Dokmanovic S, Kolovrat K, Laskaj R, Jukic V, Vrkic N, Begovac J. Effect of Extra Virgin Olive Oil on Biomarkers of Inflammation in HIV-Infected Patients: A Randomized, Crossover, Controlled Clinical Trial. Med Sci Monit. 2015 Aug 16;21:2406-13. doi: 10.12659/MSM.893881. PMID 26280823